CLINICAL TRIAL: NCT04550923
Title: Comparison of Rigid and Non-Rigid Interbody Fusion Device for Cervical Degenerative Disc Disease in Adults - A Randomized, Prospective, Multicenter Clinical Trial
Brief Title: Comparison of Rigid and Non-Rigid Interbody Fusion Device for Cervical Degenerative Disc Disease in Adults
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Baui Biotech Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202006012RIPD
Record Dates: First submitted 2020-09-02; First posted 2020-09-16 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Cervical Disc Degeneration
Keywords: Cervical Spine; Interbody Fusion; Anterior Cervical Discectomy and Fusion

STUDY DESIGN:
Intervention Model Description: Total 180 patients were enrolled, and 180 patients were randomized into either investigational device (non-rigid) group or the control (rigid) group in a 2:1 ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigational device (non-rigid) group (Experimental): Use non-rigid (Titanium Alloy, Z-Brace, Baui Biotech) interbody fusion device.
  Interventions: Combination Product: Z-Brace interbody fusion device
- Control device (rigid) group (Active Comparator): Use rigid (PEEK) interbody fusion device .
  Interventions: Combination Product: PEEK interbody fusion device

INTERVENTIONS:
Combination Product: Z-Brace interbody fusion device — Use non-rigid (Titanium Alloy, Z-Brace, Baui Biotech) interbody fusion device in Anterior Cervical Discectomy and Fusion (ACDF) surgery
  Arms: Investigational device (non-rigid) group
Combination Product: PEEK interbody fusion device — Use rigid (PEEK) interbody fusion device in Anterior Cervical Discectomy and Fusion (ACDF) surgery
  Arms: Control device (rigid) group

SUMMARY:
Rigid interbody fusion device in bulk configuration has been widely used in anterior cervical discectomy and fusion (ACDF) surgery. It is a randomized, prospective, multicenter clinical study to compare rigid and non-rigid fusion device in ACDF for cervical degenerative disc disease.

DETAILED DESCRIPTION:
This study is a randomized, prospective, multicenter clinical trial comparing rigid (PEEK) interbody fusion device with non-rigid (Titanium Alloy, Z-Brace, Baui Biotech) interbody fusion device in ACDF surgery at 11 clinical sites. ACDF was performed with stand-alone interbody fusion device and artificial bone graft (hydroxyapatite/tricalcium phosphate). Patients have 1-level or 2-level cervical degenerative disc disease approved for ACDF surgery by National Health Insurance, which is the blind, third-party, administrative approved and insurance reimbursement for surgical indication. Total 180 patients were enrolled, and 180 patients were randomized into either investigational device (non-rigid) group or the control (rigid) group in a 2:1 ratio. After confirming a patient's eligibility and having the patient sign an informed consent form, the site investigator or study coordinator call the coordinator at National Taiwan University Hospital for the randomization. Each patient will be then assigned to 1 of the treatment group according to a randomized schedule. Patient were evaluated preoperatively, one month postoperatively, and 3, 6, 12, 18, and 24 months postoperatively. Measured outcomes included overall success, Neck Disability Index (NDI), VAS neck and arm pain, adjacent range of motion, patient satisfaction, anxiety score, SF-12 MCS/PCS, major complications, subsequent surgery rate, and subsidence and fusion rate on radiological examinations. The primary endpoint was a FDA composite definition of success comprising clinical improvement and absence of major complications and secondary surgery events.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20 - 69 years;
2. Symptomatic cervical degenerative disc disease in one or two levels between C3-7 with radiculopathy or myeloradiculopathy and/or decrease muscle strength and/or abnormal sensation and/or abnormal reflexes;
3. Deficit confirmed by CT, MRI, or X-ray;
4. NDI Score of ≥ 30/100;
5. Unresponsive to non-operative treatment of at least 6 weeks or presence of progressive symptoms or signs of nerve root/spinal cord compression despite continued non-operative treatment;
6. No prior surgical procedures at the operative level and non-prior fusions at any cervical level;
7. Physically and mentally able and willing to comply with the protocol;
8. Signed informed consent;

Exclusion Criteria:

1. Patient does not meet the indication of Anterior Cervical Discectomy and Fusion (ACDF), which is under the surveillance. (Surgical indication of ACDF is approved by National Health Insurance Administration Ministry of Health and Welfare, a blinded third-party authority).
2. More than two vertebral levels required surgery;
3. Immobile levels between C1 and C7 from any cause;
4. Any prior surgery at the operative level or any prior fusion at any cervical level;
5. T-score less than -1.5 (osteoporosis evaluation)
6. Paget's disease, osteomalacia, or any other metabolic bone disease other than osteoporosis;
7. Active infection of surgical site or history of anticipated treatment for systemic infection including HIV
8. Active malignancy: a history of any invasive malignancy (except carcinoma in situ and non-melanoma skin cancer), unless treated with curative intent with no clinical signs or symptoms of malignancy in the past 5 years;
9. Marked instability of the cervical spine on resting lateral or flexion-extension radiographs;
10. Known allergy to device materials including titanium or polyetheretherketone (PEEK);
11. Segmental kyphosis of greater than 11 degrees at treatment or adjacent levels
12. Rheumatoid arthritis, lupus, or other autoimmune disease;
13. Any diseases or conditions that would preclude accurate clinical evaluation;
14. Daily, high-dose oral and/or inhaled steroid or a history of chronic use of high dose steroids;
15. Body Mass Index (BMI) > 35
16. Smoking more than one pack of cigarettes per day;

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-12-03 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline postoperative condition (if patients have major complications) | Patient were evaluated one month postoperatively, and 3, 6, 12, 18, and 24 months postoperatively.
  No adverse events (AEs) classified as major complications by Research Ethics Committee.
Change from baseline postoperative condition (if patients have subsequent surgeries) | Patient were evaluated one month postoperatively, and 3, 6, 12, 18, and 24 months postoperatively.
  No subsequent surgical intervention.
Change from baseline Subsidence and Fusion rate | Patient were evaluated one month postoperatively, and 3, 6, 12, 18, and 24 months postoperatively.
  Subsidence and fusion rate on radiological.
Change from baseline Adjacent range of motion | Patient were evaluated preoperatively, one month postoperatively, and 3, 6, 12, 18, and 24 months postoperatively.
  Adjacent range of motion on radiological.
Change from baseline Neck Disability Index (NDI) | Patient were evaluated preoperatively, one month postoperatively, and 3, 6, 12, 18, and 24 months postoperatively.
  An improvement in Neck Disability Index (NDI) score of at least 30 points for a patient with a preoperative NDI score of 60 or greater; or an improvement of at least 50% of preoperative NDI score for patients with a preoperative score of less than 60.

SECONDARY OUTCOMES:
Visual analogue scale (neck and arm and chest pain) | Patient were evaluated preoperatively, one month postoperatively, and 3, 6, 12, 18, and 24 months postoperatively.
  Patient will be evaluated by Visual analogue scale(VAS) for their neck, arm and chest pain.
  The minimum value is 0 and the maximum value is 10. Higher score means a worse outcome.
Patient Satisfaction Questionnaire | Patient were evaluated one month postoperatively, and 3, 6, 12, 18, and 24 months postoperatively.
  Patients will be surveyed by Patient Satisfaction Questionnaire. There are two questions on the questionnaire to evaluate if they are satisfied with their treatment and if they will recommend their respective surgery to a friend.
Anxiety score | Patient were evaluated preoperatively, one month postoperatively, and 3, 6, 12, 18, and 24 months postoperatively.
  The Beck Anxiety Inventory (BAI). The minimum value is 0 and the maximum value is 63. Higher scores mean a worse outcome.
Short form-12 mental component scale and physical component scale (SF-12 MCS/PCS) score | Patient were evaluated preoperatively, one month postoperatively, and 3, 6, 12, 18, and 24 months postoperatively.
  Short form-12 mental component scale and physical component scale. The minimum value of physical component scale (PCS-12) is 18.4 and the maximum value of PCS-12 is 57.8. The minimum value of mental component scale (MCS-12) is 18.7 and the maximum value of MCS-12 is 65.2. Higher scores mean a better outcome.
Number of days using Non-steroidal anti-inflammatory analgesics(NSAIDs) | Patient were evaluated preoperatively, one month postoperatively, and 3, 6, 12, 18, and 24 months postoperatively.
  Number of days using Non-steroidal anti-inflammatory analgesics(NSAIDs)
Depression Score | Patient were evaluated preoperatively, one month postoperatively, and 3, 6, 12, 18, and 24 months postoperatively.
  Beck Depression Inventory(BDI). The minimum value is 0 and the maximum value is 63. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (13):
- Taiwan (13):
  - Chung Shan Medical University Hospital, Taichung, South Dist.
  - Fu Jen Catholic University Hospital, New Taipei City, Taishan District
  - Taipei Municipal Wan Fang Hospital, Taipei, Wenshan Dist.
  - National Taiwan University Hospital Yunlin Branch, Douliu, Yunlin County
  - Taipei Medical University-Shuang Ho Hospital,Ministry of Health and Welfare, New Taipei City, Zhonghe District
  - MacKay Memorial Hospital, Taipei, Zhongshan
  - National Taiwan University Hospital, Taipei, Zhongzheng Dist.
  - National Taiwan University Hospital Hsin-Chu Branch, Hsinchu
  - China Medical University Hospital, Taichung
  - Jen-Ai Hospital Dali Branch, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Min-Sheng General Hospital, Taoyuan District
  - Chang Gung Memorial Hospital, Taoyuan District

REFERENCES:
- [Background] Zdeblick TA, Phillips FM. Interbody cage devices. Spine (Phila Pa 1976). 2003 Aug 1;28(15 Suppl):S2-7. doi: 10.1097/01.BRS.0000076841.93570.78. PMID 12897467
- [Background] Brodke DS, Zdeblick TA. Modified Smith-Robinson procedure for anterior cervical discectomy and fusion. Spine (Phila Pa 1976). 1992 Oct;17(10 Suppl):S427-30. doi: 10.1097/00007632-199210001-00014. PMID 1440038
- [Background] Shriver MF, Lewis DJ, Kshettry VR, Rosenbaum BP, Benzel EC, Mroz TE. Pseudoarthrosis rates in anterior cervical discectomy and fusion: a meta-analysis. Spine J. 2015 Sep 1;15(9):2016-27. doi: 10.1016/j.spinee.2015.05.010. Epub 2015 May 15. PMID 25982430
- [Background] Bohlman HH, Emery SE, Goodfellow DB, Jones PK. Robinson anterior cervical discectomy and arthrodesis for cervical radiculopathy. Long-term follow-up of one hundred and twenty-two patients. J Bone Joint Surg Am. 1993 Sep;75(9):1298-307. doi: 10.2106/00004623-199309000-00005. PMID 8408151
- [Background] Sugawara T, Itoh Y, Hirano Y, Higashiyama N, Mizoi K. Long term outcome and adjacent disc degeneration after anterior cervical discectomy and fusion with titanium cylindrical cages. Acta Neurochir (Wien). 2009 Apr;151(4):303-9; discussion 309. doi: 10.1007/s00701-009-0217-5. Epub 2009 Mar 5. PMID 19262984
- [Background] Elsawaf A, Mastronardi L, Roperto R, Bozzao A, Caroli M, Ferrante L. Effect of cervical dynamics on adjacent segment degeneration after anterior cervical fusion with cages. Neurosurg Rev. 2009 Apr;32(2):215-24; discussion 224. doi: 10.1007/s10143-008-0164-2. Epub 2008 Oct 10. PMID 18846395
- [Background] Barsa P, Suchomel P. Factors affecting sagittal malalignment due to cage subsidence in standalone cage assisted anterior cervical fusion. Eur Spine J. 2007 Sep;16(9):1395-400. doi: 10.1007/s00586-006-0284-8. Epub 2007 Jan 13. PMID 17221174
- [Background] Goffin J, Geusens E, Vantomme N, Quintens E, Waerzeggers Y, Depreitere B, Van Calenbergh F, van Loon J. Long-term follow-up after interbody fusion of the cervical spine. J Spinal Disord Tech. 2004 Apr;17(2):79-85. doi: 10.1097/00024720-200404000-00001. PMID 15260088
- [Background] Maiman DJ, Kumaresan S, Yoganandan N, Pintar FA. Biomechanical effect of anterior cervical spine fusion on adjacent segments. Biomed Mater Eng. 1999;9(1):27-38. PMID 10436851
- [Background] Gore DR, Gardner GM, Sepic SB, Murray MP. Roentgenographic findings following anterior cervical fusion. Skeletal Radiol. 1986;15(7):556-9. doi: 10.1007/BF00361055. PMID 3775422
- [Background] Gao X, Yang Y, Liu H, Meng Y, Zeng J, Wu T, Hong Y. A Comparison of Cervical Disc Arthroplasty and Anterior Cervical Discectomy and Fusion in Patients with Two-Level Cervical Degenerative Disc Disease: 5-Year Follow-Up Results. World Neurosurg. 2019 Feb;122:e1083-e1089. doi: 10.1016/j.wneu.2018.10.231. Epub 2018 Nov 9. PMID 30415055
- [Background] Ma Z, Ma X, Yang H, Guan X, Li X. Anterior cervical discectomy and fusion versus cervical arthroplasty for the management of cervical spondylosis: a meta-analysis. Eur Spine J. 2017 Apr;26(4):998-1008. doi: 10.1007/s00586-016-4779-7. Epub 2016 Oct 22. PMID 27771787
- [Background] Kuang L, Chen Y, Wang B, Li L, Lu G. Cervical Disk Arthroplasty Versus Anterior Cervical Decompression and Fusion for the Treatment of 2-Level Cervical Spondylopathy: A Systematic Review and Meta-analysis. Clin Spine Surg. 2016 Nov;29(9):372-382. doi: 10.1097/BSD.0000000000000395. PMID 27295435
- [Background] Hu Y, Lv G, Ren S, Johansen D. Mid- to Long-Term Outcomes of Cervical Disc Arthroplasty versus Anterior Cervical Discectomy and Fusion for Treatment of Symptomatic Cervical Disc Disease: A Systematic Review and Meta-Analysis of Eight Prospective Randomized Controlled Trials. PLoS One. 2016 Feb 12;11(2):e0149312. doi: 10.1371/journal.pone.0149312. eCollection 2016. PMID 26872258
- [Background] Ding D, Shaffrey ME. Cervical disk arthroplasty: patient selection. Clin Neurosurg. 2012;59:91-7. doi: 10.1227/NEU.0b013e31826b6fbe. No abstract available. PMID 22960519
- [Background] Jaramillo-de la Torre JJ, Grauer JN, Yue JJ. Update on cervical disc arthroplasty: where are we and where are we going? Curr Rev Musculoskelet Med. 2008 Jun;1(2):124-30. doi: 10.1007/s12178-008-9019-2. PMID 19468885
- [Background] Tahal D, Madhavan K, Chieng LO, Ghobrial GM, Wang MY. Metals in Spine. World Neurosurg. 2017 Apr;100:619-627. doi: 10.1016/j.wneu.2016.12.105. Epub 2017 Jan 3. PMID 28057595
- [Background] Epstein NE. A Review of Complication Rates for Anterior Cervical Diskectomy and Fusion (ACDF). Surg Neurol Int. 2019 Jun 7;10:100. doi: 10.25259/SNI-191-2019. eCollection 2019. PMID 31528438
- [Background] Goffin J, Casey A, Kehr P, Liebig K, Lind B, Logroscino C, Pointillart V, Van Calenbergh F, van Loon J. Preliminary clinical experience with the Bryan Cervical Disc Prosthesis. Neurosurgery. 2002 Sep;51(3):840-5; discussion 845-7. doi: 10.1227/00006123-200209000-00048. PMID 12188968
- See also: W. Bonfield MW, K.E. Tanner. Interfaces in analogue biomaterials. Acta Materialia. 1998;46（7）:2509-18. — https://doi.org/10.1016/S1359-6454(98)80035-9
- See also: Liu JT, Chen WC, Wei HW. Biomechanical evaluation of a dynamic fusion cage design for cervical spine: A finite element study. Advances in Mechanical Engineering. 2017;9（3）:1-7. — https://doi.org/10.1177/1687814017698881